CLINICAL TRIAL: NCT06685874
Title: Interstitial Lung Disease Exacerbations Study
Acronym: INDEX
Status: Active, not recruiting | Type: Observational
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University Hospitals, Leicester (Other); Nottingham University Hospitals NHS Trust (Other); North Bristol NHS Trust (Other); Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2501703
Record Dates: First submitted 2024-10-30; First posted 2024-11-13 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: Interstitial Lung Disease (ILD); Pulmonary Fibrosis
Keywords: Interstitial lung disease; Exacerbation
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with exacerbation of fibrotic interstitial lung disease: Patients with exacerbation of fibrotic interstitial lung disease as per inclusion and exclusion criteria

SUMMARY:
Interstitial lung disease (ILD) is an umbrella term covering numerous conditions that affect the lung tissue, interfering with the ability of the lungs to take up oxygen. Most ILDs get worse gradually, but sometimes patients can experience a sudden worsening in their symptoms called an acute exacerbation (AE-ILD). Most studies in this area have been done in AEs of idiopathic pulmonary fibrosis (AE-IPF), as IPF is the commonest form of ILD. AE-IPF has very poor outcomes, however AEs of other ILDs are less well studied. Furthermore, there is currently no treatment guideline or established standard of care for the management of patients with AE-fILD.

The aim of this research project is to gain a better understanding of AE-ILD in a real-world population. By looking at the clinical records of patients with AE-ILD, the study aims to describe the patient population that gets AE-ILD and how these patients are treated in the "real world" setting. The study will also gather information on patient characteristics such as type of ILD and test results at the time of AE-ILD, and see if any of these factors are associated with better/ worse outcomes in AE-ILD. Finally, the study will collect data on the treatment approaches taken, including both medical therapy such as steroid treatment, as well as specialist care team input. This data on treatment will be used to identify associations between individual treatments and outcomes, as well as to evaluate the NHS services being provided to patients with AE-ILD.

Overall, this study will enhance understanding of AE-ILD. This study will provide information to help design clinical trials to test treatments for AE-ILD, to help us create evidence-based clinical guidelines for AE-ILD, and improve the management of patients with AE-ILD.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) and other progressive fibrotic interstitial lung diseases (PF-ILDs) are increasingly common fatal disorders with a median life expectancy from diagnosis of 3-5 years. Fibrotic interstitial lung disease (fILD) is a general term for a group of conditions that involve scarring of the lung (fibrosis) with or without evidence of inflammation. While different ILDs are associated with different aetiological factors and disease courses, there is considerable overlap in the characteristics of these conditions. In general, fILDs usually progress in terms of symptoms, lung function, and radiological features, resulting in increasing symptoms and respiratory failure.

In addition to the gradual progression that is typical of fILD, these conditions can become acutely worse during episodes of acute exacerbation (AE-fILD). An AE can be defined as an acute (less than one month) deterioration in symptoms associated with new ground glass changes on CT chest and not explained by other pathology such as pulmonary embolus, pneumothorax, or cardiac failure (adapted from the definition by Collard et al for AE-IPF). The prognosis of acute exacerbations of idiopathic pulmonary fibrosis (IPF), the commonest form of fILD, is very poor (over 90% in-hospital mortality in some reports). However, there has been very little research on AEs in non-IPF fILD.

Furthermore, there is currently no treatment guideline or established standard of care for the management of patients with AE-fILD. Other significant gaps in the literature in this area, include:

* What is the typical clinical course and outcome of acute exacerbations in non-IPF fILD?
* What features predict the risk of in-hospital and post-discharge mortality from AE-fILD (e.g. age, sex, baseline diagnosis)?
* Are currently used treatments for AE-fILD effective? How should AE-fILD be managed (steroids, oxygen therapy etc)?
* How well are aspects of care that patients find important (e.g. provision of specialist palliative care, opportunities to discuss advanced care planning, and oxygen therapy) delivered to patients with AE-fILD?

There are significant gaps in the literature in the field of AE-fILD. Much of the current practice in AE-fILD management is based on clinical judgement, and adequately powered randomised controlled trials to identify appropriate treatment approaches have not been performed. This has led to significant heterogeneity in the approach to AE-fILD between clinicians and centres, an issue illustrated by the fact that only one of seven NHS trusts in the East Midlands has a treatment guideline specific for the management of AE-fILD (unpublished data). This lack of consistency in approach poses a significant challenge to the design of randomised control trials, as heterogeneity within a standard care control arm can obscure any specific signals. Furthermore, in the absence of RCTs, there is the potential that clinicians may unintentionally use interventions that are harmful.

The study is an observational cohort study of patients admitted to hospital with AE-fILD to answer the questions listed above. These data will help to clarify research priorities in this area, and identify areas where care could improve and allow us to make recommendations for clinical care. The study will also use these data to inform and generate hypotheses for future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to an acute NHS trust during study period 1st September 2022-31st August 2023 with an underlying or new diagnosis of an ILD (defined by ICD-10 codes in Table 1) with a fibrotic phenotype (established fibrosis on current or previous radiological imaging) AND
* Increasing pulmonary symptoms AND
* No extra-parenchymal cause identified as primary cause of admission

  * Segmental or larger pulmonary embolus as main discharge diagnosis in absence of acute exacerbation features on imaging
  * Pleural effusion as main discharge diagnosis
  * Pneumothorax as main discharge diagnosis in absence of acute exacerbation features on imaging
  * Left sided heart failure or volume overload

Exclusion Criteria

* No underlying or new diagnosis of ILD with a fibrotic phenotype
* Acute presentation of pneumonitis/ILD without evidence of fibrosis (Table 2)
* Non-respiratory related hospital admission (no increasing pulmonary symptoms)
* Respiratory related hospital admission due to extra-parenchymal cause

  * Segmental or larger pulmonary embolus as main discharge diagnosis in absence of acute exacerbation features on imaging
  * Pleural effusion as main discharge diagnosis
  * Pneumothorax as main discharge diagnosis in absence of acute exacerbation features on imaging
  * Left sided heart failure or volume overload
* Participant signatory to NHS National Data Opt Out
* Elective/non-emergency admission
* Admission under non-medical specialty
* In cases where there are >=1 eligible admissions only the first (index) admission shall be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with fibrotic interstitial lung disease admitted to hospital with exacerbation of pulmonary fibrosis as per inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Transplant free survival | 90 days post date of hospital admission
  Transplant-free survival

SECONDARY OUTCOMES:
Transplant free survival | Date of discharge from hospital for index admission (Up to 24 hours), 30 days, 90 days (Primary endpoint), 6 months, 1 year
  Transplant free survival
Pulmonary Function Testing | 6 months and 12 months from date of index admission
  Change in forced vital capacity (FVC) from pre-admission values
Pulmonary function testing | 6 months and 12 months from date of index admission
  Change in diffusion capacity (DLCO) from pre-admission values
Oxygen | At the point of discharge from index admission (up to 24 hours)
  Use of long term or ambulatory oxygen

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gibbons, MBChB, Principal Investigator — Royal Devon and University healthcare trust
Locations (3):
- United Kingdom (3):
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - North Bristol NHS Trust, Bristol
  - Royal Devon University Hospitals NHS Foundation Trust, Exeter

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to lack of informed consent.